CLINICAL TRIAL: NCT02267434
Title: A Randomized, Placebo-controlled, Parallel Group, Patient-blinded, Multi-center, Phase I Pilot Study to Assess Tolerability and Safety of Two Doses of AFFITOPE® PD03A Formulated With Adjuvant to Patients With Early Parkinson's Disease
Brief Title: Study Assessing Tolerability and Safety of AFFITOPE® PD03A in Patients With Early Parkinson's Disease
Acronym: AFF011
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affiris AG (Industry)
Collaborators: PROSENEX AmbulatoriumbetriebsGMBH (Unknown); Medical University Innsbruck (Other); Forschungszentrum Juelich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFFiRiS 011; 2014-000568-16 (EudraCT Number)
Record Dates: First submitted 2014-09-04; First posted 2014-10-17 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Parkinson Disease; Neurodegenerative Diseases
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose AFFITOPE® PD03A + Adjuvant (Experimental): 4 injections of 15µg AFFITOPE® PD03A/ adjuvanted, once every 4 weeks
  1 boost immunization 36 weeks after first injection
  Interventions: Biological: Low dose AFFITOPE® PD03A + Adjuvant
- High dose AFFITOPE® PD03A + Adjuvant (Experimental): 4 injections of 75µg AFFITOPE® PD03A/ adjuvanted, once every 4 weeks
  1 boost immunization 36 weeks after first injection
  Interventions: Biological: High dose AFFITOPE® PD03A + Adjuvant
- Adjuvant without active component (Placebo Comparator): 4 injections of Placebo once every 4 weeks
  1 administration 36 weeks after first injection
  Interventions: Biological: Adjuvant without active component

INTERVENTIONS:
Biological: Low dose AFFITOPE® PD03A + Adjuvant — s.c. injection
  Arms: Low dose AFFITOPE® PD03A + Adjuvant
Biological: High dose AFFITOPE® PD03A + Adjuvant — s.c. injection
  Arms: High dose AFFITOPE® PD03A + Adjuvant
Biological: Adjuvant without active component — s.c. injection
  Arms: Adjuvant without active component

SUMMARY:
Study AFF011 is a randomized controlled parallel Group phase I study to investigate the safety and tolerability of two doses of the vaccine AFFITOPE® PD03A given to patients with early Parkinson's disease.

In total 36 patients will be enrolled in 3 independent groups (2 treatment groups, 1 Placebo group), each consisting of 12 patients. The patients will be randomized to either receive 15µg or 75µg AFFITOPE® PD03A formulated with adjuvant or the reference substance without active component (Placebo). Over a study duration of 52 weeks, the study participants receive 4 injections as basic immunization in a 4-weekly interval and 1 boost immunization 36 weeks after the first injection. Male and female patients aged 45 to 70 years can participate in the trial. 2 study sites in Austria (Innsbruck and Vienna) will be involved.

AFF011 is part of a project SYMPATH funded by the European Commission (FP7-HEALTH-2013-INNOVATION-1 project; N° HEALTH-F4-2013-602999).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with IPS diagnosed for less than 4 years and who present in Hoehn & Yahr Stages I/II and fulfill the United Kingdom Parkinson's Disease Society Brain Bank Criteria
* The result of a DAT-SPECT and MRI examination of the patient's brain has to be consistent with the diagnosis of PD
* Written Informed Consent Form signed and dated by the patient
* Age between 45 and 70
* Female patients of childbearing potential are eligible if they use a medically accepted contraceptive method
* A potential participant treated with conventional PD therapies must be on stable doses for at least 3 months prior to Visit 0 and during the entire trial period and must be a stable responder
* Accepted PD medications include the following: levodopa (alone or in combination with benserazide, carbidopa), Catechol-O-methyltransferase inhibitors (entacapone, tolcapone), amantadine, non-ergot dopamine agonists (pramipexol, ropinirol, rotigotine), monoamine oxidase-B inhibitors (rasagiline, selegiline) and anticholinergic medication
* A potential participant has to be on stable doses of all medications he/she is taking because of consisting illnesses according to medical history (except PD therapies, these will be recorded separately) for at least 30 days prior to Visit 0, if considered relevant by the PI
* Upon PI's opinion, no visual or auditory impairments that would reduce the patients' ability to complete study questionnaires or be unable to receive instructions for these

Exclusion Criteria:

* Pregnant women
* Sexually active women of childbearing potential who are not using a medically accepted birth control method throughout the study
* Participation in another clinical trial within 3 months before Visit 0
* History of questionable compliance to visit schedule; patients not expected to complete the clinical trial
* Presence or history of allergy to components of the vaccine, if considered relevant by the PI
* Contraindication for MRI imaging such as metallic endoprosthesis or stent implantation in the last 6 months or allergy to MRI contrast agent
* Contraindication for DAT-SPECT
* Contraindication for lumbar puncture such as anticoagulation
* Dementia
* History and/or presence of autoimmune disease, if considered relevant by the PI
* Recent (≤3 years since last specific treatment) history of cancer (Exceptions: basal cell carcinoma, intraepithelial cervical neoplasia)
* Active infectious disease (e.g., Hepatitis B, C)
* Presence and/or history of Immunodeficiency (e.g., HIV)
* Significant systemic illness (e.g., chronic renal failure, chronic liver disease, poorly controlled diabetes, poorly controlled congestive heart failure, other deficiencies), if considered relevant by the PI
* History of significant psychiatric illness such as schizophrenia, bipolar affective disorder or psychotic depression
* Parkinson-like disease secondary to drug therapy side effects (e.g., due to exposure to medications that deplete dopamine [reserpine, tetrabenazine] or block dopamine receptors [neuroleptics, antiemetics]
* Parkinson-plus syndromes (e.g. MSA, PSP)
* Heredodegenerative disorders
* Alcoholism or substance abuse within the past year (alcohol or drug intoxication)
* Prior and/or current treatment with experimental immunotherapeutics including intravenous immunoglobulin
* Prior and/or current treatment with immunosuppressive drugs
* Change in dose of standard treatments for PD within 3 months prior to Visit 0
* Change in dose of previous and current medications which the patient is taking because of consisting illnesses according medical history (except PD therapies, these will be recorded separately) within the last 30 days prior to Visit 0, if clinically relevant
* Treatment with deep brain stimulation
* Venous status rendering it impossible to place an i.v. access
* L-Dopa related motor complications (response fluctuations and/or dyskinesia)
* Evidence for genetic forms of PD: leucine-rich repeat kinase 2 and Parkin

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of patients who withdraw due to Adverse Events (AEs) | 12 months
  The withdrawal criteria (continuation decision) in regards to the number of patients who withdraw due to AEs as well as the reason for withdrawal will be evaluated.
Occurrence of Adverse Events and Serious Adverse Events | 12 months
  Evaluation of Adverse Events and Serious Adverse Events in regards to autoimmune reactions
New findings or Change in pre-existing findings assessed in physical and neurological examinations over time (study period) | 12 months
Change in vital signs and Body mass over time (study period) | 12 months
  The Evaluation of vital signs includes the changes in blood pressure, heart rate, respiratory rate and Body temperature over time (measured at each visit).
Safety related Evaluation of MRI results of patients' brain after visit 5 and visit 8 compared to baseline | 12 months
  MRI safety measures will e.g. include the occurrence of inflammatory reactions (meningoencephalitis), new/changed hemorrhages and lacunar infarcts.
Clinical significance/changes in laboratory parameters over time (study period) | 12 months
  Laboratory assessment includes hematology, biochemistry, coagulation, serology and urinanalysis.

SECONDARY OUTCOMES:
Immunological activity of AFFITOPE® vaccine PD03A | 12 months
  Titer of vaccination induced antibodies directed towards vaccine components, alpha- and beta synuclein
Change in motor symptoms at visit 8 and visit 11 compared to baseline | 12 months
  Change in motor symptoms: MDS Unified Parkinson's Disease Rating Scale (UPDRS) II and III
Change in non-motor symptoms at visit 8 and visit 11 compared to baseline | 12 months
  Change in non-motor symptoms: PDQ-39 (Parkinson's Disease Quality of Life-39)/PD non-motor symptom score, MDS UPDRS I (Movement Disorder Society Unified Parkinson's Disease Rating scale), cognitive test battery, HAM-D (Hamilton Depression Rating Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Werner Poewe, MD, Principal Investigator — Medical University Innsbruck, Department of Neurology, Innsbruck 6020, Austria
Locations (2):
- Austria (2):
  - Medical University Innsbruck, Department of Neurology, Innsbruck
  - Studienzentrum der PROSENEX, AmbulatoriumbetriebsgesmbH an der Confraternität -Privatklinik Josefstadt, Vienna